CLINICAL TRIAL: NCT06036407
Title: Improving Access to Screening for Hearing Loss After Childhood Cancer - a Novel Community-based Approach
Brief Title: Screening for Hearing Loss After Childhood Cancer
Acronym: HEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Krebsforschung Schweiz, Bern, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SCCSS_Ototox
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Childhood Cancer; Hearing Loss
Keywords: Ototoxicity; Late Effect; Ototoxic; Follow-up care; Screening
MeSH Terms: conditions — Neoplasms; Hearing Loss; Ototoxicity | interventions — Hearing Tests

STUDY DESIGN:
Masking Description: All participants undergo a hearing test (intervention).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Participants (Experimental): Participants make an appointment at a hearing aid shop in Switzerland. They get the results right after the hearing test and may take it to their respective physician if wanted.
  Interventions: Diagnostic Test: Hearing test

INTERVENTIONS:
Diagnostic Test: Hearing test — Participants visit a local hearing aid shop to assess their hearing function
  Other Names: Hearing evaluation; Hearing assessment; Hearing screening

SUMMARY:
The HEAR-study pilots and evaluates a national, low-threshold screening program to detect hearing problems in Swiss adult childhood cancer survivors.

Participants will conduct a hearing test in a local hearing aid shop and report about their experiences at the shop in questionnaires and interviews. The screening program will be evaluated using the RE-AIM framework.

DETAILED DESCRIPTION:
Hearing loss is an adverse event in childhood cancer survivors (CCS). It is caused by ototoxic cancer treatments, in particular platinum chemotherapy, cranial radiation with doses of ≥30 Gray, and surgery involving the auditory system.

Undetected hearing loss, even if mild, can have a strong impact on life. It affects language acquisition in infants, school performance and communication, thus interfering with survivors' professional life, social integration, and quality of life. Although hearing loss is irreversible in most CCS, it can be treated with speech therapy or hearing aids; therefore, early detection is important. Unfortunately, one third of CCS in Switzerland with ototoxic treatment did not get auditory follow-up screening after completion of acute cancer treatment.

CCS in follow-up care are often discharged to primary care, particularly for late effects that are not life threatening such as hearing loss. Multidisciplinary follow-up clinics for adult CCS were recently initiated in Switzerland. These provide risk-adapted individual examinations and counseling for CCS by organizing several medical examinations within one or two days, but capacity is limited. Additionally, extended visits in large hospitals are costly for the healthcare system and time-consuming for CCS. Low-threshold screening programs that are easily accessible and less time-consuming might therefore be a valuable addition to improve screening for hearing loss among CCS.

The main rationale for this study is to test a novel community-based, low-threshold screening approach for hearing loss in CCS in Switzerland. The screening program is tested and evaluated using the RE-AIM (reach, effectiveness, adoption, implementation, maintenance) framework for assessing health interventions including reach, effectiveness, adoption, implementation and maintenance (see outcome measures). The second aim is to use the data obtained to close knowledge gaps on risk factors of ototoxicity after childhood cancer. This will eventually lead to improved care and higher quality of life for affected CCS.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with childhood cancer according to the international classification of childhood cancer, edition 3 (ICCC3) main groups
* Diagnosed before the age 21
* Diagnosed in Switzerland
* Registered in the Swiss Childhood Cancer Registry
* Recovered & survived ≥2 years after diagnosis
* Diagnosed between 1976-2019
* Treated in one of the clinics of the Swiss Paediatric Oncology Group
* Exposed to any chemotherapy and/or radiation to the head, neck or spine (TBI included)
* Written informed consent

Exclusion Criteria:

* Recently contacted for other studies (January 2022-July 2022)
* Not German/French speaking
* No postal address available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 476 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Reach: Number/proportion of written informed consents | 1 day after signed informed consent is sent back
  Reach measures to which extent the target population participates in the program by assessing representativeness and participant population coverage.
  Number of written informed consents is counted and divided by the number of people invited to get the response rate.
Reach: Number/proportion of participants that consented, who participated in screening program (i.e. completed hearing test) | 4 weeks after participant completed hearing test
  Number of participants that conducted hearing test is counted and divided by the number of people that consented to participate in the screening program.
Reach: Comparing characteristics of (non-)responders | 1 day after signed informed consent is sent back
  Characteristics of responders (signed informed consent) are compared to those of non-responders. Data from the childhood cancer registry on age at study, age at diagnosis, diagnosis, treatment regimens and urbanicity are extracted and compared by using cross-field tabulations and chi-square tests for categorical variables and independent sample t-tests and analysis of variance for continuous variables.
  This comparison gives information on the representativeness of the study population.
Reach: Motives for participation | 3 months after participant completed hearing test
  Motives for participation are assessed through interviews with study participants after the hearing test. They are asked why they participated.
Effectiveness: Number/proportion of participants with (newly) detected hearing loss | 4 weeks after participant completed hearing test
  Effectiveness focuses on evaluating immediate and long-term impacts (positive and negative) of the intervention. It examines whether the intervention achieves its objectives (i.e., detecting hearing loss) and what other impacts it might have (e.g. mental health).
  Participants fill out two follow-up questionnaires 4 weeks after the hearing test and 6 months after the hearing test. In the first follow-up questionnaire, participants are asked what the result of the hearing test was. This data is compared to a baseline data that is collected through a questionnaire before the hearing test. Numbers of hearing impaired persons at baseline and at follow up are then compared.
Effectiveness: Number/proportion of participants with (newly) detected hearing loss who contacted their treating healthcare professional. | 6 months after participant completed hearing test
  In the second follow-up questionnaire, participants are asked, if they consulted a physician after receiving their hearing test result and if they have done something about their hearing impairment (if present). These numbers give information on the impact of the screening program on the population (e.g. new hearing aids).
Effectiveness: Other possible effects on mental health (newly detected hearing loss, reminded of disease) | 3 months after participant completed hearing test
  In the interviews with study participants after the hearing test, they are asked how they felt before, during and after the hearing test and if something changed in their lifes since they got their hearing test results.
  Emerging topics are collected, analysed and integrated in the second follow-up questionnaire to get more information from more participants.
Adoption: Satisfaction, opinions and suggestions of participants and key stakeholders | 3 months after participant completed hearing test
  Adoption assesses how the program is adopted by target settings (i.e., hearing aid shops, health care professionals), assessing stakeholder's willingness/readiness to adopt and implement the intervention.
  In interviews with study participants, they are asked about their experiences with the screening program, how it compared to existing follow-up care programs, its advantages and disadvantages and their overall opinions on the program.
  To get insight from all stakeholders involved, acousticians from the hearing aid shops and health care professionals from the fields of pediatric oncology, follow-up care and/or audiology are also interrogated.
  Acousticians and health care professionals are asked for their opinions on the program and suggestions for improvement. Further, they are asked for challenges or difficulties they encountered or anticipated.
Adoption: Geographical distribution of hearing aid shops visited during the study | 4 weeks after participant completed hearing test
  To get insight on how the program was used by the study population, observational data from the hearing aid provider are collected to see where the participants visited the hearing aid shops.
Implementation: Fidelity and consistency to the intervention protocol. | Six months after hearing test
  Implementation evaluates the feasibility of implementing the intervention within real-world contexts, assessing the extent to which the intervention is delivered consistently and as intended. It also includes required resources.
  In the interviews with acousticians, they are asked about their experiences with study participants during the hearing test. They are asked if study participants differ from usual customers and in what way and if they treated them differently than usual customers (i.e. find out if they changed protocol in some way).
  Further, they are asked if they reached capacity limits in their respective hearing aid shops and if they needed additional resources (than usual).
  These interviews inform the design of a questionnaire to all acousticians that performed hearing tests on a study participant to get more information from more persons.
Implementation: Estimated costs for implementation | Six months after hearing test
  Costs for implementation are calculated based on empirical values and data from the hearing aid shops: Work time, infrastructure, skills, expertises.
Maintenance: Opinions of stakeholders and participants on the continuation of the screening program | Six months after participant conducted hearing test
  Maintenance investigates the possibility of continuing the program beyond the research project, considering its long-term sustainability.
  Assessed through interviews with and questionnaires to participants and stakeholders:
  * Opinions of stakeholders and participants on the continuation of the screening program
  * Identification of necessary requirements and resources for the program's future continuation
  * Potential integration of the program into the existing follow-up care programs for childhood cancer survivors

SECONDARY OUTCOMES:
Assessing hearing function in childhood cancer survivors | Examinations (hearing tests) between July 2022 and July 2023
  Audiograms of adult CCS in Switzerland are collected from the hearing tests. The hearing function is then assessed using the International Society of Paediatric Oncology (SIOP) Boston Ototoxicity Scale for grading hearing loss.
Identify risk factors for hearing loss in CCS | Hearing test results between July 2022 and July 2023
  Data from the childhood cancer registry on age at study, age at diagnosis, diagnosis, treatment regimens as well as from questionnaires (environmental risk factors) are extracted and used to identify risk factors associated with hearing loss.
  Risk factors are identified by calculating Odds Ratios using univariable and multivariable logistic regression.

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Kuehni, MD, Principal Investigator — Institute of Social and Preventive Medicine, University of Bern
Locations (1):
- Institute for Social and Preventive Medicine, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiss A, Sommer G, Kasteler R, Scheinemann K, Grotzer M, Kompis M, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Long-term auditory complications after childhood cancer: A report from the Swiss Childhood Cancer Survivor Study. Pediatr Blood Cancer. 2017 Feb;64(2):364-373. doi: 10.1002/pbc.26212. Epub 2016 Sep 21. PMID 27650356
- [Background] Clemens E, van den Heuvel-Eibrink MM, Mulder RL, Kremer LCM, Hudson MM, Skinner R, Constine LS, Bass JK, Kuehni CE, Langer T, van Dalen EC, Bardi E, Bonne NX, Brock PR, Brooks B, Carleton B, Caron E, Chang KW, Johnston K, Knight K, Nathan PC, Orgel E, Prasad PK, Rottenberg J, Scheinemann K, de Vries ACH, Walwyn T, Weiss A, Am Zehnhoff-Dinnesen A, Cohn RJ, Landier W; International Guideline Harmonization Group ototoxicity group. Recommendations for ototoxicity surveillance for childhood, adolescent, and young adult cancer survivors: a report from the International Late Effects of Childhood Cancer Guideline Harmonization Group in collaboration with the PanCare Consortium. Lancet Oncol. 2019 Jan;20(1):e29-e41. doi: 10.1016/S1470-2045(18)30858-1. PMID 30614474
- [Background] Bass JK, Liu W, Banerjee P, Brinkman TM, Mulrooney DA, Gajjar A, Pappo AS, Merchant TE, Armstrong GT, Srivastava D, Robison LL, Hudson MM, Krull KR. Association of Hearing Impairment With Neurocognition in Survivors of Childhood Cancer. JAMA Oncol. 2020 Sep 1;6(9):1363-1371. doi: 10.1001/jamaoncol.2020.2822. PMID 32729886
- [Background] Weiss A, Sommer G, Schindera C, Wengenroth L, Karow A, Diezi M, Michel G, Kuehni CE; Swiss Paediatric Oncology Group (SPOG). Hearing loss and quality of life in survivors of paediatric CNS tumours and other cancers. Qual Life Res. 2019 Feb;28(2):515-521. doi: 10.1007/s11136-018-2021-2. Epub 2018 Oct 10. PMID 30306534
- [Background] Khairi Md Daud M, Noor RM, Rahman NA, Sidek DS, Mohamad A. The effect of mild hearing loss on academic performance in primary school children. Int J Pediatr Otorhinolaryngol. 2010 Jan;74(1):67-70. doi: 10.1016/j.ijporl.2009.10.013. Epub 2009 Nov 12. PMID 19913305
- [Background] Weiss A, Kuonen R, Brockmeier H, Grotzer M, Candreia C, Maire R, Senn P, Stieger C, Rosenfeld J, Veraguth D, Kompis M, Scheinemann K, Kuehni CE; Swiss Pediatric Oncology Group (SPOG). Audiological monitoring in Swiss childhood cancer patients. Pediatr Blood Cancer. 2018 Mar;65(3). doi: 10.1002/pbc.26877. Epub 2017 Dec 12. PMID 29230928
- [Background] Babecoff S, Mermillod F, Marino D, Gayet-Ageron A, Ansari M, Fernandez E, Gumy-Pause F. Long-term follow-up for childhood cancer survivors: the Geneva experience. Swiss Med Wkly. 2022 Apr 7;152:w30153. doi: 10.4414/smw.2022.w30153. eCollection 2022 Mar 28. PMID 35429234
- [Background] Michel G, Kuehni CE, Rebholz CE, Zimmermann K, Eiser C, Rueegg CS, von der Weid NX; Swiss Paediatric Oncology Group (SPOG). Can health beliefs help in explaining attendance to follow-up care? The Swiss childhood cancer survivor study. Psychooncology. 2011 Oct;20(10):1034-43. doi: 10.1002/pon.1823. Epub 2010 Aug 4. PMID 20687196
- [Background] Michel G, Gianinazzi ME, Eiser C, Bergstraesser E, Vetsch J, von der Weid N, Kuehni CE; Swiss Paediatric Oncology Group. Preferences for long-term follow-up care in childhood cancer survivors. Eur J Cancer Care (Engl). 2016 Nov;25(6):1024-1033. doi: 10.1111/ecc.12560. Epub 2016 Aug 23. PMID 27550385
- [Result] Jorger P, Nigg C, Mader L, Strebel S, Kompis M, Tomasikova Z, Schindera C, Michel G, von der Weid NX, Ansari M, Waespe N, Kuehni CE. A Health Service Research Study on a Low-Threshold Hearing Screening Program for Childhood Cancer Survivors in Switzerland: Protocol for the HEAR Study. JMIR Res Protoc. 2025 May 21;14:e63627. doi: 10.2196/63627. PMID 40397950
- [Result] Jorger P, Nigg C, Zarkovic M, Sommer G, Kompis M, Michel G, Ansari M, Waespe N, Kuehni CE. Awareness about the risk of hearing loss after ototoxic treatments in Swiss childhood cancer survivors. Patient Educ Couns. 2025 Jul;136:108764. doi: 10.1016/j.pec.2025.108764. Epub 2025 Mar 27. PMID 40179545
- See also: Study protocol of the HEAR-study — https://preprints.jmir.org/preprint/63627
- See also: A Health Service Research Study on a Low-Threshold Hearing Screening Program for Childhood Cancer Survivors in Switzerland: Protocol for the HEAR Study — https://www.researchprotocols.org/2025/1/e63627/authors